CLINICAL TRIAL: NCT03051438
Title: The Feasibility and Advantages of Subxiphoid Uniportal Video-assisted Thoracoscopic Surgery in Pulmonary Lobectomy.A Retrospective Study
Brief Title: The Feasibility and Advantages of Subxiphoid Uniportal Video-assisted Thoracoscopic Surgery in Pulmonary Lobectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Xueying Yang (Other)
Responsible Party: Sponsor-Investigator, Xueying Yang, Professor, Shengjing Hospital
Organization: Shengjing Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: B451-1
Record Dates: First submitted 2017-02-07; First posted 2017-02-13 (Actual); Last update posted 2018-05-24 (Actual); Status verified 2018-05

CONDITIONS: Lobectomy; Subxiphoid Uniportal Video-assisted Thoracoscopic Surgery

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Subxiphoid uniportal VATS (Other): retrospectively analyzed and compared perioperative data for patients who underwent subxiphoid uniportal and traditional three-port VATS lobectomies
  Interventions: Procedure: Subxiphoid uniportal VATS
- Three-port VATS (Other): retrospectively analyzed and compared perioperative data for patients who underwent subxiphoid uniportal and traditional three-port VATS lobectomies
  Interventions: Procedure: Three-port VATS

INTERVENTIONS:
Procedure: Subxiphoid uniportal VATS — Patients were placed in a supine position, and the operating table was manipulated as needed to elevate the appropriate side of the body for surgery. The surgical procedures followed principles of pulmonary resections; in particular, similar to mediastinal lymphadenectomy for lung cancer, these procedures involved the individual dissection of veins, arteries and lobar bronchi.
  Arms: Subxiphoid uniportal VATS
Procedure: Three-port VATS — The surgical procedures followed principles of pulmonary resections; in particular, similar to mediastinal lymphadenectomy for lung cancer, these procedures involved the individual dissection of veins, arteries and lobar bronchi
  Arms: Three-port VATS

SUMMARY:
Uniportal video-assisted thoracoscopic surgery (VATS) lobectomy has emerged as a promising and exciting approach for minimally invasive thoracic surgery. However, nearly all reported uniportal VATS lobectomies have been performed via the intercostal route, and chest wall trauma has still occurred. Here,the investigators undertook novel uniportal VATS technique involving a subxiphoid route for pulmonary lobectomies to evaluate the feasibility and advantages.

ELIGIBILITY:
Inclusion Criteria:

* Patients with lung cancer can be undertook the subxiphoid uniportal VATS or three-port VATS

Exclusion Criteria:

* Contraindications in patients with lung cancer

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 86 (Estimated)
Dates: Start 2016-01 (Actual); Primary Completion 2018-06 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With Abnormal Laboratory Values and/or Adverse Events That Are Related to Treatment | 17 months

CONTACTS AND LOCATIONS:
Locations (1):
- Shengjing Hospital, Shenyang, Liaoning, China

REFERENCES:
- [Result] Liu CC, Wang BY, Shih CS, Lin WC. Subxyphoid single-incision thoracoscopic pulmonary metastasectomy. Thorac Cancer. 2015 Mar;6(2):230-2. doi: 10.1111/1759-7714.12189. Epub 2015 Mar 2. PMID 26273365
- [Result] Liu CY, Lin CS, Liu CC. Subxiphoid single-incision thoracoscopic surgery for bilateral primary spontaneous pneumothorax. Wideochir Inne Tech Maloinwazyjne. 2015 Apr;10(1):125-8. doi: 10.5114/wiitm.2015.48572. Epub 2015 Jan 27. PMID 25960803
- [Result] Gonzalez-Rivas D, Yang Y, Lei J, Hernandez L, Jiang G. Subxiphoid uniportal video-assisted thoracoscopic middle lobectomy and anterior anatomic segmentectomy (S3). J Thorac Dis. 2016 Mar;8(3):540-3. doi: 10.21037/jtd.2016.02.63. PMID 27076952
- [Result] Hernandez-Arenas LA, Lin L, Yang Y, Liu M, Guido W, Gonzalez-Rivas D, Jiang G, Jiang L. Initial experience in uniportal subxiphoid video-assisted thoracoscopic surgery for major lung resections. Eur J Cardiothorac Surg. 2016 Dec;50(6):1060-1066. doi: 10.1093/ejcts/ezw189. Epub 2016 Jul 11. PMID 27401700
- [Result] Song N, Zhao DP, Jiang L, Bao Y, Jiang GN, Zhu YM, Ding JA. Subxiphoid uniportal video-assisted thoracoscopic surgery (VATS) for lobectomy: a report of 105 cases. J Thorac Dis. 2016 Mar;8(Suppl 3):S251-7. doi: 10.3978/j.issn.2072-1439.2016.02.32. PMID 27014471
- [Result] Liu CC, Wang BY, Shih CS, Liu YH. Subxiphoid single-incision thoracoscopic left upper lobectomy. J Thorac Cardiovasc Surg. 2014 Dec;148(6):3250-1. doi: 10.1016/j.jtcvs.2014.08.033. Epub 2014 Aug 23. No abstract available. PMID 25240526
- [Derived] Yang X, Wang L, Zhang C, Zhao D, Lu Y, Wang Z. The Feasibility and Advantages of Subxiphoid Uniportal Video-Assisted Thoracoscopic Surgery in Pulmonary Lobectomy. World J Surg. 2019 Jul;43(7):1841-1849. doi: 10.1007/s00268-019-04948-6. PMID 31065773